CLINICAL TRIAL: NCT05872490
Title: Predictive Factors Associated With Continued Driving in Old Age : a Mixed Methods Approach
Brief Title: Predictors Associated With Maintaining Driving in Old Age
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Gerontopole Auvergne Rhone-Alpes (AURA) (Other); Jean Monnet University (Other); University Hospital, Lille (Other); Centre de Recherche Hospitalier Universitaire de Marseille (Unknown)
Responsible Party: Principal Investigator, Nathalie BARTH, Project leader, Sociologist, Centre Hospitalier Universitaire de Saint Etienne
Other Study IDs: GA-2021-06
Record Dates: First submitted 2023-05-10; First posted 2023-05-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Aged, 80 and Over
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Older 80 people: Semi-structured interviews were conducted for the qualitative research. In addition, a driving habits questionnaire was administered. To complete this questionnaire, medical data from the PROOF cohort were collected.The PROOF cohort is a prospective study for which enrollment began in 2001. The main objective is to evaluate the predictive value of Autonomic Nervous System (ANS) activity and its decline during follow-up on the occurrence of serious and cerebral events, and on all-cause mortality, in a general population of subjects of homogeneous age. Participants were included in the study if they were 65 years of age (plus or minus 2 years) at the time of inclusion and registered on the electoral list of the city of St Etienne, had not had a previous myocardial infarction or stroke and were non-insulin dependent.
  Interventions: Other: Semi-structured interviews; Other: Questionnaire
- Attending physicians: Semi-structured interviews were conducted for the qualitative research
  Interventions: Other: Semi-structured interviews
- law enforcement: Semi-structured interviews were conducted for the qualitative research
  Interventions: Other: Semi-structured interviews
- certified driver's license physicians: Semi-structured interviews were conducted for the qualitative research
  Interventions: Other: Semi-structured interviews
- geriatricians: Semi-structured interviews were conducted for the qualitative research
  Interventions: Other: Semi-structured interviews
- driving instructors: Semi-structured interviews were conducted for the qualitative research
  Interventions: Other: Semi-structured interviews
- personal assistance services: Semi-structured interviews were conducted for the qualitative research
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — An interview guide was developed for each population. Depending on the population interviewed, this interview guide focuses on the current state of driving, the obstacles and levers to driving, the representations related to driving by the elderly, their opinion concerning the implementation of a potential aptitude test and more generally their opinion on policies related to road safety.
Other: Questionnaire — The questionnaire asks people aged 80 and over included in the PROOF cohort about their relationship to driving, their driving status, their societal and personal environment, the circumstances in which they stopped driving, recent accidents and, more generally, their driving habits.
  Groups: Older 80 people

SUMMARY:
The goal of this observational study is to learn about predictors associated with maintaining driving in old age. The main questions it aims to answer are :

* which and how medical factors can influence stopping or maintaining driving (quantitative research)
* how social environment can influence stopping or maintaining driving (quantitative research)
* what are the needs of all the actors in the field (qualitative research)
* know about the opinions and practices of all the actors in the field (qualitative research) Participants will be ask to answer questions in an interview taking about an hour. Quantitative research will ask participants to fill out a questionnaire about social environment.

DETAILED DESCRIPTION:
FAMACO is a project led by Gérontopôle Auvergne Rhône-Alpes (AURA) and Chaire Santé des Ainés of the Jean Monet University, supported by the Observatoire National Interministériel de la Sécurité Routière (ONISR), that aims prevent the loss of autonomy of the elderly population by identifying predictors associated with maintaining driving in old age. This is a mixed quantitative and qualitative prospective study.

Quantitative study identify medical factors linked to stopping driving by analysis data from "PROnostic of factors OF cardiovascular or neurovascular disease" (PROOF) cohort. In addition, a questionnaire on the social environment was addressed to participants.

Qualitative study focus on identifying the expectations and needs of all concern populations : elderly divers, elderly former drivers, general practitioner, geriatrician, certified driver's license physician, law enforcement, driving instructors and emergency services. This qualitative study will be carried out on three different sites : Saint-Etienne, Marseille, and Lille.

ELIGIBILITY:
Inclusion criteria :

* being part of one of the population studied (older 65 people ; attending physicians ; law enforcement ; certified driver's license ; physicians ; geriatricians ; driving instructors ; personal assistance services)
* live in Saint-Etienne, Marseille or Lille

Exclusion criteria :

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 7 populations are included in the study: older 65 people ; attending physicians ; law enforcement ; certified driver's license ; physicians ; geriatricians ; driving instructors ; personal assistance services. For each of them, the respondents are based in one of the three investigation sites: Saint-Etienne, Lille or Marseille. For people aged 65 and over, a questionnaire is also distributed.
Sampling Method: Non-Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Views and representations of the different populations on the conduct of the elderly | Day 1
  Representations and habits of elderly driving were study by individual semi-directive interviews. The aims is to identify, in the accounts of experiences, the practices, the relationship to driving and to other forms of transport, the lived experience, the representations of driving and ageing.

SECONDARY OUTCOMES:
Driving habits of elderly | Day 1
  Habits of elderly driving were study by a questionnaire to understand the social and personal environment in relation to driving habits.
  The Evaluation of Precariousness and health Inequalities in health Examination Centers Score (EPICES score) was measured in this questionnaire. This individual indicator allows for the measurement of precariousness by taking into account its multidimensional nature.The questionnaire is composed of 11 questions which summarise 90% of the precariousness situation of a subject. Each question is assigned a coefficient and the sum of the answers gives the score. The score is continuous and varies from 0 (no insecurity) to 100 (maximum insecurity). The threshold of 30 is considered as the threshold of precariousness.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BARTH, PhD, Study Chair — GERONTOPOLE AURA
Locations (3):
- France (3):
  - Nathalie Barth, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - François Puisieux, Lille
  - Sylvie Bonin-Guillaume, Marseille